CLINICAL TRIAL: NCT01283347
Title: Phase II Study of 18F-DTBZ: The Differential Diagnosis of Parkinson's Disease and Monitoring the Severity of Disease by VMAT2 PET Imaging
Brief Title: 18F-DTBZ for l Diagnosis of Parkinson's Disease and Monitoring the Severity of Disease by VMAT2 PET Imaging
Acronym: 8F-DTBZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, NJI90OKM, Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 98-2160A
Record Dates: First submitted 2011-01-11; First posted 2011-01-26 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-DTBZ for Parkinson's Disease (Experimental): 25 age-matched healthy volunteers will be enrolled. For assessing the correlation between the 18F-DTBZ binding and the severity of disease, the patients with PD will be divided into three groups according to their motor scores: mild, moderate, and advanced. We will enroll 25 patients in each group. Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping, each subject will have 3 visits in this study, as one screening visit, one imaging visit, and one safety evaluation visit.
  Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.
  Interventions: Drug: 18F-DTBZ

INTERVENTIONS:
Drug: 18F-DTBZ — During this study, subjects will receive a single i.v. administration of approximately 10 mCi 18F-FP-(+)-DTBZ immediately prior to imaging.
  The proposed dose for this study is based on our phase I study. At the proposed human dose of 10 mCi, the whole body effective dose (ED) will be approximately 680 mrem. The estimated human ED is expected to be comparable to or below the range of other approved brain imaging agents, such as 18F-FDG

SUMMARY:
The primary objective of this protocol is to analyze the sensitivity and specificity of 18F-DTBZ PET to the differential diagnosis of Parkinson's Disease (PD) and normality. Secondary, the investigators will analyze the correlation between the 18F-DTBZ binding and the severity of disease of PD and the role of 18F-DTBZ PET in the monitoring disease severity.

DETAILED DESCRIPTION:
25 age-matched healthy volunteers will be enrolled. For assessing the correlation between the 18F-DTBZ binding and the severity of disease, the patients with PD will be divided into three groups according to their motor scores: mild, moderate, and advanced. We will enroll 25 patients in each group. Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping, each subject will have 3 visits in this study, as one screening visit, one imaging visit, and one safety evaluation visit.

Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders and 50~80 years old.
2. Written and dated informed consent by self or by legal representative, to be obtained before any of the study procedures
3. Healthy male or female subjects with no evidence of significant neurologic impairment by history.
4. Seventy-five PD subjects will be divided as three subgroups according to the severity of disease: mild (Modified Hoehn and Yahr stage 1 to 2), moderate (Modified Hoehn and Yahr stage 2.5 to 3), and advanced (Modified Hoehn and Yahr stage 4 to 5).
5. All the PD subjects should be fulfilled the UK Parkinson's Disease Society Brain Bank criteria of "possible" or "probable" PD. The age of disease onset should be older than 50 years.

Exclusion Criteria:

1. Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
2. Any subject who has a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.
3. History of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
4. History or presence of QTc prolongation.
5. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
6. Any documented abnormality in the brain by CT or MRI of brain, which might contribute to the motor function, such as hydrocephalus, multiple infarction and encephalomalacia, will be excluded. Mild cortical atrophy and non-specific white matter changes will be allowed.
7. Patients who have the evidence of secondary

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the sensitivity and specificity of 18F-DTBZ PET to the differential diagnosis of PD and normality for drug safety assessment | 2 year
  To evaluate the sensitivity and specificity of 18F-DTBZ PET to the differential diagnosis of PD and normality.
  During this study, subjects will receive a single i.v. administration of approximately 10 mCi 18F-FP-(+)-DTBZ immediately prior to imaging

SECONDARY OUTCOMES:
To analyze the correlation between the regionally reduced 18F-DTBZ binding and the severity of disease of PD. | 1 years
  The objectives of this study is to determine the sensitivity and specificity of 18F-DTBZ PET to the differential diagnosis of PD and normality, and to analyze the correlation between the regionally reduced 18F-DTBZ binding and the severity of disease of PD

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Song Lu, Principal Investigator — Department of Neurological ,LIN KOU
Locations (1):
- Chang Gung Memory Hpspital, Taoyuan District, Taiwan